CLINICAL TRIAL: NCT02677753
Title: InterStim Implantation Rates Following Percutaneous Nerve Evaluation With Fluoroscopy Versus Without
Brief Title: Percutaneous Nerve Evaluation With Fluoroscopy Versus Without
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Sean Francis, Principal investigator, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15.0034
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Overactive Bladder; Urinary Incontinence; Fecal Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence; Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluoroscopy guided PNE (Active Comparator): Fluoroscopy will be utilized to assist with placement and/or confirm correct placement of lead wires.
  Interventions: Radiation: Fluoroscopy
- PNE without fluoroscopic guidance (No Intervention): No fluoroscopy will be used during or after the placement of the lead wires.

INTERVENTIONS:
Radiation: Fluoroscopy
  Arms: Fluoroscopy guided PNE

SUMMARY:
The investigators propose a randomized control trial comparing the rate of implantation of the InterStim device following Percutaneous Nerve Evaluation (PNE) performed with or without fluoroscopic guidance.

DETAILED DESCRIPTION:
Sacral nerve stimulation (SNS) is a well-established treatment for refractory urinary urgency, frequency, retention and urge incontinence as well as fecal incontinence. Patients whose symptoms are refractory to more conservative therapies such as behavioral modification and/or medications are candidates for SNS. The InterStim system consists of a permanent tined lead and implantable pulse generator (IPG) or battery that delivers the sacral neuromodulation. This device is typically implanted after patients have a successful response to a trial of sacral neuromodulation with a temporary lead and external battery. The temporary lead placement is known as a Percutaneous Nerve Evaluation (PNE) and is typically done in as an outpatient procedure using local anesthetic. It is standard practice to use fluoroscopy intraoperatively to confirm correct placement of the permanent lead. Additionally, some physicians also use fluoroscopy to confirm correct placement of temporary lead during PNE while others place the lead based on anatomical landmarks and expected elicited responses for S3 stimulation.

The investigators propose a randomized control trial comparing the rate of implantation of the InterStim device following (PNE) performed with or without fluoroscopic guidance.

ELIGIBILITY:
Inclusion Criteria:

* Women age >18
* English speakers
* Patients with urinary urgency, frequency, or urge incontinence refractory to at least 1 other intervention who elect to undergo PNE

Exclusion Criteria:

* Patients in whom bilateral leads cannot be placed
* Pregnant women
* Prisoners
* Less than 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean L Francis, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Physicians, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
* Age
  * Race
  * BMI
  * Preoperative diagnosis
  * Previous treatments for urinary urgency, frequency, retention, and/or urinary or fecal incontinence
  * Percent improvement in symptoms as determined by pre and post PNE voiding diaries
  * Whether or not InterStim implanted within 3 months of PNE
  * Date of PNE

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluoroscopy Guided PNE: Fluoroscopy will be utilized to assist with placement and/or confirm correct placement of lead wires.
  Fluoroscopy
Period: Overall Study
Arm/Group | Fluoroscopy Guided PNE | PNE Without Fluoroscopic Guidance
Started | 37 | 38
Completed | 36 | 38
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoroscopy Guided PNE | PNE Without Fluoroscopic Guidance | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.94 (14.29) | 57.84 (14.01) | 57.89 (14.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian participants | 29 | 35 | 64
Indication for PNE, Urge urinary incontinence [Count of Participants; unit: Participants] | 30 | 33 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With InterStim Implantation Following PNE With or Without Use of Fluoroscopy
Description: Percentage of PNEs that have permanent neuromodulation device implanted by 3 months
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fluoroscopy Guided PNE | PNE Without Fluoroscopic Guidance
Number analyzed (Participants) | 36 | 38
Participants | 21 | 18

ADVERSE EVENTS:
Time Frame: Within 3 months after PNE placement
Description: Patients were queried at time of procedure as well as post op and adverse events were recorded. The PI also reviewed the charts at completion of study and collected any additional adverse event data
Arm/Group | Fluoroscopy Guided PNE | PNE Without Fluoroscopic Guidance
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/38
Other Adverse Events (participants affected / at risk) | 5/36 | 3/38
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoroscopy Guided PNE (N=36) | PNE Without Fluoroscopic Guidance (N=38)
Pain, premature of retained lead (Renal and urinary disorders) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There were no sponsors for this study

DOCUMENTS (2):
  • Informed Consent Form (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT02677753/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT02677753/Prot_SAP_001.pdf